CLINICAL TRIAL: NCT05954546
Title: Overall Survival (OS) in Patients With Metastatic BRAFV600-mutant Melanoma Treated With Encorafenib Plus Binimetinib in the COLUMBUS Trial Versus in Real-world Practice Data
Brief Title: A Study to Compare How Effective is Encorafenib Plus Binimetinib in Real-world and Clinical Trial Settings
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C4221035
Record Dates: First submitted 2023-07-12; First posted 2023-07-20 (Actual); Results first posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Drug: Enco+bini — Patients with BRAF mutant + receiving encorafenib and binimetinib combination treatment

SUMMARY:
Brief summary The purpose of this study is to compare how effective, encorafenib plus binimetinib is in the real-world and clinical trial settings. And produce results to show that combining data on encorafenib plus binimetinib from both the real-world and clinical trial settings is possible for future research studies.

This study group is identified from the database who:

* Have taken at least 1 order or administration of encorafenib plus binimetinib treatment after the confirmation of having metastatic melanoma after 27 June 2018.
* Are at least 18 years of age at the time of first encorafenib plus binimetinib initiation (index date).
* Had never received encorafenib plus binimetinib or had received first-line immunotherapy at the start of the study.
* Have ECOG status of 0 or 1 at the index date.
* have available data on the number of deaths in an area or group of people.

Patients will be followed from the date that the patient started the first encorafenib plus binimetinib treatment (treatment initiation) up to their last date of data availability. Last date of data availability could be the date of following events: patient lost to follow up at the clinic, death, or end of the database (January 2020). The database timeframe is June 2018 to January 2020.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of melanoma (International Classification of Diseases 9th or 10th Revision Clinical Modification - ICD-9-CM: 172.X; ICD-10-CM: C43.x) and secondary malignancy or metastasis (ICD-9-CM: 196.x, 197.x, 198.x; ICD-10-CM: C77.x, C78.x, C79.x).
* Confirmed BRAF V600E/V600K activating mutation reported in the data based on laboratory or genetic analysis results.
* At least 1 order or administration of ENCO+BINI treatment

Exclusion criteria:

* Patients without information on mortality
* Patients with ECOG performance status ≥ 2 (at the time of randomization for patients from COLUMBUS, during the baseline period for patients in Flatiron Electronic Health Record)
* Patients with a history of or concurrent uveal or mucosal melanoma, basal cell or squamous cell carcinoma (as per trial inclusion criteria); this exclusion will also be applied to RWD patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with BRAF mutant + metastatic melanoma receiving encorafenib and binimetinib
Sampling Method: Non-Probability Sample
Enrollment: 275 (Actual)
Dates: Start 2023-07-21 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4221035

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data of eligible participants with v-Raf murine sarcoma viral oncogene homolog B protein (BRAF) V-600 mutant melanoma who aged greater than or equal to 18 years at the time of initiating treatment with Encorafenib plus Binimetinib (ENCO+BINI) was collected retrospectively.
Pre-assignment Details: Data sources: COLUMBUS trial (NCT01909453) and Flatiron Health Electronic Health Records (EHR) real-world database (RWD). Planned cohorts in this study: 1) ENCO+BINI, clinical trial data (CTD) from COLUMBUS; 2) ENCO+BINI (RWD) from Flatiron EHR. Available retrospective data was evaluated in this observational study from 21-Jul-2023 to 31-Dec-2023 [approximately 5.35 months].
Groups:
- Encorafenib+Binimetinib (CTD): Participants with BRAFV600-mutant metastatic melanoma, who were enrolled between 30-December-2013 to 15-September-2020 in phase 3 COLUMBUS trial and treated with Encorafenib 450 mg once daily (QD) and Binimetinib 45 mg twice daily (BID) (ENCO+BINI) were included.
- Encorafenib+Binimetinib (RWD): Eligible participants with BRAFV600-mutant metastatic melanoma, identified from Flatiron Health Database between 27-June-2018 to 01-January-2022 and treated with Encorafenib 450 mg QD and Binimetinib 45 mg BID (ENCO+BINI) were included.
Period: Overall Study
Arm/Group | Encorafenib+Binimetinib (CTD) | Encorafenib+Binimetinib (RWD)
Started | 192 | 83
Completed | 192 | 83
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Eligible participants whose data was retrieved and observed in the study.
Groups:
- Encorafenib+Binimetinib (CTD): Participants with BRAFV600-mutant metastatic melanoma, who were enrolled between 30-December-2013 to 15-September-2020 in phase 3 COLUMBUS trial and treated with Encorafenib 450 mg QD and Binimetinib 45 mg BID (ENCO+BINI) were included.
- Total: Total of all reporting groups
Arm/Group | Encorafenib+Binimetinib (CTD) | Encorafenib+Binimetinib (RWD) | Total
Number analyzed (Participants) | 192 | 83 | 275
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.2 (13.6) | 60.4 (14.2) | 57.5 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 36 | 113
  Male | 115 | 47 | 162
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Here, Number analyzed signifies number of participants for whom data was collected and was available to be reported.
  Participants
    number analyzed (Participants) | 181 | 71 | 252
    White | 181 | 71 | 252

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: As per COLUMBUS trial, OS was defined as the time from the date of randomization to the date of death due to any cause; if death was not observed, participants were censored at the date of last contact or the data analysis cut-off date, whichever occurred first. As per Flatiron EHR, OS was defined as the time from the index date to the date of death; participants without a date of death were censored at their last known activity date or the end of the follow-up period, whichever occurred first. Index date in each treatment group was defined as the date of treatment initiation. Kaplan-Meier analyses was used for analysis.
Time Frame: COLUMBUS: From date of randomization until death or censoring (approx 80.5 months); Flatiron: From index date until death due or censoring or end of follow-up period (approx 42.2 months)
Population: Analysis population included all eligible participants whose data were retrieved and observed in this study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Encorafenib+Binimetinib (CTD) | Encorafenib+Binimetinib (RWD)
Number analyzed (Participants) | 192 | 83
Months | 33.6 [25.5 to 39.5] | 24.0 [16.4 to NA] — To estimate an upper limit of 95% confidence limit (CI), enough follow-up and events were required after the median OS reached. But beyond median OS, participants at risk and events were insufficient. Hence, upper limit of 95% CI could not be estimated.
Statistical Analysis 1: Comparison: Encorafenib+Binimetinib (CTD) vs Encorafenib+Binimetinib (RWD); Statistical analysis data is presented for Encorafenib+Binimetinib (RWD) relative to Encorafenib+Binimetinib (CTD) (reference); Test type: Other; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.62 to 1.72] — Hazard ratio (HR) was estimated using multivariable Cox proportional hazard models

ADVERSE EVENTS:
Time Frame: All cause mortality: COLUMBUS trial approximately 80.5 months and Flatiron EHR RWD approx 42.2 months. For adverse events it was not applicable as adverse event data was not planned to be collected.
Description: This study is retrospective, it involves data that exist as structured data by the time of study start. The minimum criteria for reporting an adverse event (AE) (i.e., identifiable participant, identifiable reporter, a suspect product, and event) cannot be met. Hence, adverse events were not planned to be collected and are not reported.
Arm/Group | Encorafenib+Binimetinib (CTD) | Encorafenib+Binimetinib (RWD)
All-Cause Mortality (participants affected / at risk) | 131/192 | 28/83
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-24): https://cdn.clinicaltrials.gov/large-docs/46/NCT05954546/Prot_SAP_000.pdf